CLINICAL TRIAL: NCT03756987
Title: Does Ultrasound-guided Erector Spinae Plane Block Improve Postoperative Quality of Recovery After Video-assisted Thoracic Surgery
Brief Title: Does ESPB Improve Postoperative Quality of Recovery After VATS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Clinical Professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K2018-10-001
Record Dates: First submitted 2018-11-13; First posted 2018-11-28 (Actual); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Postoperative Pain
Keywords: ultrasound-guided; erector spinae plane block; quality of recovery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Saline Solution; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization sequence will be computer generated. Allocation concealment will be carried out via concealed assignments in opaque, sealed, and consecutively numbered envelopes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESPB group (Experimental): Patient will receive a single shot of Ropivacaine injection 0.5% 25 mL injected at the erector spinae plane.
  Interventions: Drug: Ropivacaine Injection
- Control Group (Placebo Comparator): Patient will receive a single shot of normal saline 25 mL injected at the erector spinae plane.
  Interventions: Drug: Normal saline

INTERVENTIONS:
Drug: Ropivacaine Injection — Ropivacaine will be injected in the erector spinae plane
  Other Names: ESPB group
  Arms: ESPB group
Drug: Normal saline — Normal saline will be injected in the erector spinae plane.
  Other Names: Control group
  Arms: Control Group

SUMMARY:
Video-Assisted Thoracoscopic Surgery (VATS) is a minimally invasive surgery. Despite reduced surgical trauma compared to the traditional thoracotomy approach, pain control after VATS remains challenging. Regional analgesia may be a crucial component of multimodal postoperative pain management. The use of nerve blocks, such as the recently described erector spinae plane block (ESPB) has been shown in case reports to reduce pain and thus has the potential to improve patient recovery. This study aims to test the hypothesis that ultrasound-guided SPB would improve the quality of recovery after VATS by reducing acute postsurgical pain.

DETAILED DESCRIPTION:
VATS is a minimally invasive surgical technique to remove intrathoracic lesions. VATS has become increasingly popular and gradually becoming the standard of care for lung surgery. Although acute pain after VATS is less than the traditional thoracotomy, patients still experience moderate amount of pain within the first 24 hours. However, the optimal regional analgesic technique for VATS procedures has not been established.

Thoracic epidural analgesia (TEA) and paravertebral block (PVB) have been tried to improve postoperative analgesia after VATS. Although TEA and PVB provides superior analgesia, these technologies accompanied by the rare but serious complications involving epidural hematoma, pneumothorax and total spinal anesthesia.

Erector spinae plane block (ESPB) is a novel and simple ultrasound-guided regional anesthetic technique, providing analgesia for the ipsilateral hemithorax. Ultrasound guidance is believed to improve peripheral and regional nerve block success rates and safety. ESPB is a technically easy to perform. ESPB has only been reported in case series but so far, no adverse events such as hypotension, hematoma or infection has been reported.

Given its safety, ease of performance and efficacy, the study aims to verify the hypothesis that combines ESPB with general anesthesia would accelerate functional recovery after breast cancer surgery. Our secondary aims were to examine ESPB's effect on analgesic outcomes (e.g., postoperative pain intensity, cumulative opioid consumption, postoperative nausea and vomiting, dizziness, the postanesthesia care unit discharge time and patients' satisfaction) in patients undergoing VATS.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' physical status class of I or II
* scheduled for elective VATS

Exclusion Criteria:

* a history of allergy to local anesthetics
* known coagulation disorders
* infection near the puncture site
* chronic opioid use
* inability to communicate,
* other reasons that not appropriate for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-12-28 (Actual); Primary Completion 2019-11-12 (Actual); Study Completion 2019-11-14 (Actual)

PRIMARY OUTCOMES:
the 40-item Quality of Recovery (QoR-40) score | The QoR-40 questionnaire was completed by patients at 24 hours after surgery.
  QoR-40 incorporates 40 questions assessing 5 dimensions of recovery, including emotional status, physical comfort, psychological support, physical independence, and pain. The global QoR-40 score ranges from 40 (extremely poor quality of recovery) to 200 (excellent quality of recovery).

SECONDARY OUTCOMES:
postoperative pain: numeric rating scale | Acute postoperative pain was assessed using an numeric rating scale (NRS) at 0.5, 1, 2, 4, 8, 12, 24, and 48 hours following video-assisted thoracic surgery.
  0-10 numeric rating scale for pain (0 minimal pain and 10 worst pain ever)
cumulative opioid consumption | Up to 48 hours after surgery.
  We recorded opioid(sufentanil) consumption at 48 hours after surgery. consumption at 6, 24, and 48 hours after surgery.cumulative opioid (sufentanil) consumption
PACU discharge time | Up to 2 hours
  Post-anesthetic recovery length of stay in minutes
Incidence of nausea and vomiting | Up to 48 hours
  Patient reported sensation of nausea and incidence of vomiting related to opioid intake.
Incidence of dizziness | Up to 48 hours
  Patient reported incidence of dizziness related to opioid intake.
patient's satisfaction: numeric rating scale | Patient's satisfaction was evaluated at 48 hours postoperatively.
  Patient's satisfaction was evaluated with a 10-point numerical rating scale ranging from 1 (highly unsatisfactory) to 10 (highly satisfactory).

CONTACTS AND LOCATIONS:
Overall Officials: Xiaochun Zheng, MD, Study Director — Fujian Provincial Hospital
Locations (1):
- Yusheng Yao, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: Yes
It is not yet known if there will be a plan to make individual participant data (IPD) available.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 3 years following article publication.
Access Criteria: All of the individual participant data collected during the trial, the study protocol, statistical analysis plan, and clinical study report can be accessed with approval from the corresponding author.